CLINICAL TRIAL: NCT01847391
Title: A Phase 1, Single-Blind, Randomized, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of GS-6615 in Healthy Subjects
Brief Title: A Phase 1 Study to Assess the Safety,Tolerability, and Pharmacokinetics of GS-6615 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: GS-US-279-0102
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Ischemic Heart Disease
Keywords: Ischemic Heart Disease; Heart Disease
MeSH Terms: conditions — Myocardial Ischemia; Heart Diseases | interventions — eleclazine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Randomized to 6 mg once daily (Days 1-7) followed by 3 mg once daily (Days 8-21) of GS-6615 or matching placebo
  Interventions: Drug: GS-6615; Drug: Placebo
- Cohort 2 (Experimental): Randomized to 12 mg once daily (Days 1-7) followed by 6 mg once daily (Days 8-21) of GS-6615 or matching placebo
  Interventions: Drug: GS-6615; Drug: Placebo
- Cohort 3 (Experimental): Randomized to 20 mg once daily (Days 1-7) followed by 9 mg once daily (Days 8-21) of GS-6615 or matching placebo
  Interventions: Drug: GS-6615; Drug: Placebo

INTERVENTIONS:
Drug: GS-6615 — GS-6615 tablet(s) administered orally once daily
Drug: Placebo — Placebo tablet(s) to match GS-6615 administered orally once daily

SUMMARY:
This is a phase 1, single-blind, randomized, placebo-controlled, multiple ascending dose study aimed to assess the safety, tolerability, and pharmacokinetics of GS-6615 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Weight of at least 50 kg with body mass index (BMI) between 18 and 30 kg/m2
* Female subjects must be of non-childbearing potential as defined per the protocol
* Male subjects with female partners of childbearing potential must be using protocol acceptable methods of contraception
* Willing and able to comply with the requirements of the protocol and directions
* Willing to avoid consumption of grapefruit, grapefruit juice and Seville oranges
* Willing to avoid consumption of nicotine (including nicotine gum) and alcoholic beverages

Exclusion Criteria:

* Ongoing or history of any medical or surgical condition that, in the judgment of the Investigator, might jeopardize the subject's safety or interfere with the study objectives
* History of meningitis or encephalitis, seizures, migraines, tremors, myoclonic jerks, sleep disorder, anxiety, syncope, head injuries or a family history of seizures
* Any abnormal ECG findings, abnormal laboratory value, or physical examination findings at Screening judged to be clinically significant
* Any abnormal neurological examination findings at Screening that is judged as clinically significant
* Hemoglobin < 12 g/dL
* Serology test positive for HIV, or hepatitis B or C
* Positive urine drug test (including cotinine or ethanol)
* Use of systemic prescription medications or over the counter (OTC) medication, including multivitamins, and dietary and herbal supplement
* Use of any experimental or investigational drug or device within 30 days
* Female subjects who are of childbearing potential, pregnant or lactating
* Donation or loss of blood within 8 weeks and/or donation of plasma within 7 days
* History of drug or alcohol abuse
* Psychosocial or addictive disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GS-6615 | Up to 65 days
  The primary outcome measure is the safety and tolerability of GS-6615 including neurological findings, adverse events, clinical laboratory tests, vital signs and ECG data (PR, RR, QRS, QT, and QTc [Fridericia] interval).
Pharmacokinetic (PK) profile of GS-6615 | Up to 65 days
  The primary outcome measure is the PK profile of GS-6615 which will be measured with Cmax, Tmax, AUCtau, AUC0-∞, T1/2, CL/F, VSS/F, and R.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Layug, MD, Study Director — Gilead Sciences
Locations (1):
- Investigational Site, Madison, Wisconsin, United States